CLINICAL TRIAL: NCT05274100
Title: A Phase 1, Pharmacokinetic Comparability Study of Intravenous and Subcutaneous Administration of Risankizumab in Healthy Subjects
Brief Title: Study of Intravenous and Subcutaneous Administration of Risankizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M19-128
Record Dates: First submitted 2022-03-08; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Risankizumab; SKYRIZI
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1: Risankizumab Dose A (Experimental): Participants will receive risankizumab dose A.
  Interventions: Drug: Risankizumab
- Group 2: Risankizumab Dose B (Experimental): Participants will receive risankizumab dose B.
  Interventions: Drug: Risankizumab
- Group 3: Risankizumab Dose C (Experimental): Participants will receive risankizumab dose C.
  Interventions: Drug: Risankizumab
- Group 4: Risankizumab Dose D (Experimental): Participants will receive risankizumab dose D.
  Interventions: Drug: Risankizumab
- Group 5: Risankizumab Dose D (Experimental): Participants will receive risankizumab dose D.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection via prefilled syringe (PFS)
  Other Names: SKYRIZI
  Arms: Group 1: Risankizumab Dose A
Drug: Risankizumab — Intravenous Infusion
  Other Names: SKYRIZI
  Arms: Group 4: Risankizumab Dose D; Group 5: Risankizumab Dose D
Drug: Risankizumab — Subcutaneous Injection via on-body delivery system (OBDS)
  Other Names: SKYRIZI
  Arms: Group 2: Risankizumab Dose B; Group 3: Risankizumab Dose C

SUMMARY:
The primary objectives of this study are to assess the relative bioavailability of risankizumab in on-body delivery system (OBDS) versus the prefilled syringe (PFS) (Substudy 1) and to assess the relative bioavailability of risankizumab in the to-be-marketed Dose A liquid vial versus the Dose B liquid vial used in the Phase 3 studies (Substudy 2).

ELIGIBILITY:
Inclusion Criteria:

- Body weight less than 100.00 kg at Screening and upon initial confinement.

Exclusion Criteria:

- Previous exposure to any anti-IL-12/23 or anti-IL-23 treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Adverse Events (AEs) | Up to approximately 140 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Maximum Observed Serum Concentration (Cmax) | Up to approximately 113 days
  Maximum observed serum concentration (Cmax) of risankizumab.
Time to Cmax (Tmax) | Up to approximately 113 days
  Time to Cmax of risankizumab.
Apparent Terminal Phase Elimination Rate Constant (β) | Up to approximately 113 days
  Apparent terminal phase elimination rate constant (β) of risankizumab.
Terminal Phase Elimination Hhalf-life (t1/2) | Up to approximately 113 days
  Terminal phase elimination half-life (t1/2) of risankizumab.
Area Under Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) | Up to approximately 113 days
  AUCt of risankizumab.
AUC From Time 0 to Infinity (AUCinf) | Up to approximately 113 days
  AUCinf of risankizumab.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- United States (8):
  - Anaheim Clinical Trials LLC /ID# 222821, Anaheim, California
  - Altasciences Clinical Los Angeles, Inc /ID# 222238, Cypress, California
  - Clinical Pharmacology of Miami /ID# 225392, Miami, Florida
  - PPD Clinical Research Unit /ID# 222362, Orlando, Florida
  - Acpru /Id# 222349, Grayslake, Illinois
  - PPD Clinical Research Unit -Las Vegas /ID# 222363, Las Vegas, Nevada
  - PPD Clinical Research Unit - Austin /ID# 222361, Austin, Texas
  - Spaulding Clinical Research LLC /ID# 225405, West Bend, Wisconsin